CLINICAL TRIAL: NCT00215826
Title: A Randomized, Dose-ranging Study of Alferon® LDO {Low Dose Oral Interferon Alfa-n3 (Human Leukocyte Derived)} in Normal Volunteers and/or Asymptomatic Subjects With Exposure to a Person Known to Have SARS or Possible SARS
Brief Title: Study of Alferon® LDO (Low Dose Oral) in Normal Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIM ImmunoTech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LDO-102
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Severe Acute Respiratory Syndrome
Keywords: SARS; Alferon LDO; Low Dose Oral Interferon ALFA-n3; Human Leukocyte Derived; Exposure to SARS; Possible SARS
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 650 IU
  Interventions: Drug: Alferon LDO
- 2 (Active Comparator): 1300 IU
  Interventions: Drug: Alferon LDO

INTERVENTIONS:
Drug: Alferon LDO

SUMMARY:
The purpose of this trial is to conduct a randomized dose-ranging study to evaluate the safety and activity of orally administered low dose interferon alfa-n3 as an antiviral and immunomodulator in asymptomatic subjects with recent exposure to a person with severe acute respiratory syndrome (SARS) or possible SARS. The primary objective of this pilot study is to determine an Alferon LDO dose level that increases or upregulates genes known to be mediators of interferon response. Secondary endpoints include the development of SARS symptomatology, rate of hospitalization, and mortality rate. In the event that no subjects with recent exposure to a person with SARS or possible SARS are available, this study will be conducted with 10 normal volunteers.

DETAILED DESCRIPTION:
This study will be an open-label, randomized, outpatient study in subjects potentially infected with the SARS-CoV (SARS-associated coronavirus) or normal volunteers using two dose levels of LDO interferon.

Subjects will be randomized to receive Alferon® LDO (natural interferon alfa-n3) in a buffer solution once each day for 10 consecutive days at doses equal to 650 IU or 1300 IU/day.

Pretherapy baseline evaluations will be performed prior to randomization.

Subjects will be randomly assigned to each dose level, and both dosage levels will be started concurrently. Drug will be dispensed for a ten day treatment period, during which time any clinical symptoms and adverse events will be evaluated. Laboratory samples (2.5 ml blood) for microarray analysis evaluations will be made twice during baseline and 12-14 hours following doses 1, 5, and 10 on study days 2, 6, and 11, respectively.

The conduct of this study will comply with International Conference on Harmonisation - Good Clinical Practice (ICH - GCP) and the 1996 or later version of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years of age.
2. Asymptomatic with close contact within the last 5 days with a person known to have possible SARS (SARS RUI-2 (SARS Report under investigation), RUI-3, RUI-4) or probable SARS or confirmed SARS using the Centers for Disease Control and Prevention (CDC) Supplement B: SARS Surveillance, Appendix B1: Revised Council of State and Territorial Epidemiologists (CSTE) SARS Surveillance Case Definition (Attachment II).
3. Oral temperature < 100.4°F (<38°C)
4. Subjects must be asymptomatic with regard to SARS related clinical symptoms including any signs of a respiratory illness.
5. Serum creatinine ≤ 1.5 x ULN (upper limit of normal); serum bilirubin ≤ 1.5 x ULN.
6. Total white blood cells (WBC) ≥ 3000/mm3, platelet count ≥ 100,000/mm3 and granulocytes ≥ 1500 mm3.
7. Hemoglobin > 10.0 g/dl.
8. ALT (alanine aminotransferase) and AST (aspartate aminotransferase) < 4 times upper normal limit.
9. C-reactive protein serum level in normal range
10. Serum albumin > 2.0 g/dl.
11. Written informed consent.
12. Females must either be of non-child bearing potential, or utilize an effective form of contraception and have a negative pregnancy test prior to randomization.

Exclusion Criteria:

1. Pregnant or nursing women, or women not using an effective form of contraception.
2. Less than 18 years of age.
3. Active intravenous (IV) drug users.
4. Receipt of any immunosuppressive agent, chemotherapy, or systemic steroids within 45 days of study entry.
5. Receipt of any immunomodulator such as BCG (bacille Calmette Guerin) vaccine, isoprinosine, or similar experimental agents within 45 days of study entry.
6. Evidence of HIV or other viral infections including chronic hepatitis, or other active gastrointestinal, renal, respiratory, endocrine, hematologic, cardiovascular, neurological, or psychiatric disorder that would limit the subject's ability to complete the study period.
7. Unlikely or unable to comply with the requirements of the protocol.
8. Patients unwilling or unable to give informed consent.
9. Patients on any other concurrent experimental medication.
10. Patients using any form of interferon therapy during the 6 weeks prior to study entry.
11. Hospitalized subjects, or those with an active viral infection other than possible SARS, within 2 weeks of study entry.
12. Transfusion dependent subjects (subjects requiring > 1 unit of packed RBC [red blood cells] per month within the 3 months prior to study entry).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-11; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Gene expression analysis | Days 0, 2, 6, 11, 12, 15, 20 and 40
  Increased expression of genes known to be mediators of interferon response.

SECONDARY OUTCOMES:
SARS CoV Antibody | Days 0, 15, 20 and 40
  Development of clinical SARS-CoV symptomatology
SARS-CoV infection
  Hospitalization for SARS-CoV infection and Death

CONTACTS AND LOCATIONS:
Overall Officials: Tommy R. Tong, M.D., Principal Investigator — The Kowloon West Cluster Clinical Research Ethics Committee
Locations (1):
- Princess Margaret Hospital, Lai Chi Kok, Kowloon, Hong Kong